CLINICAL TRIAL: NCT05506865
Title: Efficacy and Safety of Indacaterol vs Tiotropium From Baseline to 24 Weeks, in Women With Moderate-severe COPD Secondary to Biomass Exposure: Randomized, Non Inferior, Open Label, Parallel Groups Clinical Trial
Brief Title: Efficacy and Safety of Indacaterol vs Tiotropium in Women With COPD Secondary to Biomass Exposure
Acronym: EMERALD2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Respiratory Diseases, Mexico (Other Government)
Responsible Party: Principal Investigator, Alejandra Ramirez Venegas, Principal Investigator, National Institute of Respiratory Diseases, Mexico
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: C 26-12
Record Dates: First submitted 2022-07-06; First posted 2022-08-18 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2022-09

CONDITIONS: COPD
Keywords: COPD; Biomass
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Indacaterol (Experimental): Indacaterol 150 mcgr, one inhaled capsule, dose once daily, with dry powder inhaler device.
  Interventions: Drug: Indacaterol
- Tiotropium (Active Comparator): Tiotropium 18 mcgr, 1 inhaled capsule, dose once daily, with dry powder inhaler device
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: Indacaterol — Indacaterol, one inhales capsule, 150 mcgr, by dry powder dispositive
  Other Names: Onbrize
  Arms: Indacaterol
Drug: Tiotropium — Tiotropium 18 mcgr, one inhaled capsule, by dry powder inhaler handihaler
  Other Names: Spiriva
  Arms: Tiotropium

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a disease that produces a high rate of social and economic health mortality and morbidity not only in our country but in the international field. The causes of this disease are well-known, being smoking what produces the major portion and the less (but no less important) frequently, biomass exposure (when people cook or warm the house). It is described that the COPD secondary to biomass exposure it is approximately a third half of all the cases in cohorts in patients with this disease.

Patients clinical affection with COPD by biomass is different from the one described in patients by smoking, being the most frequent the affection peripheral airway, with major proportion of symptoms such as dyspnoea, cough and expectoration (Phenotype "chronic bronchitis"), major frequency of exacerbations, as well as, major affection in the quality of life related to health and a minimum emphysema proportion.

Currently, there is a trend of paying attention on the outcomes based on patients, such as symptoms, quality of life and the risk prevention (exacerbations) as it is exposed in the strategy GOLD 2011. In that way, the bronchodilators use as a pillar in the COPD due to the utility for the exacerbation prevention, symptomatic improvement and in quality of life, predominating the utility of ultra long-acting bronchodilators, such as tiotropium. Recently, it is available more information on new bronchodilators as indacaterol, demonstrating at least no inferiority effect on FEV1, inspiring capacity (in fact, discreet superiority on the last one) and symptoms. A functional outcome clinically important is the capacity of exercising; Six-Minute Walk Test (6MWT) has been widely used to predict prognosis of COPD secondary to smoking. This test has not been evaluated in predicting the response to the specific treatment in patients with COPD secondary to biomass exposure.

Long-acting bronchodilators have been demonstrated a benefit to the patients with COPD by smoking, in the exercising capacity measured by 6MWT. There are several reasons why this outcome could be more relevant especially in this population: inhabit in rural areas where people walk long distances, most of them are women and they are usually in charge of all the housework.

Almost all the studies reported until now exclude patients with COPD due to some cause other than smoking. Due to the lack of information on this item and the particularities in this clinical and functional characteristics observed in this kind of patients, it is considered that these patients will be benefit with the use of ultra long-acting bronchodilators, to long period and, potentially can be observed additional benefits in the decrease of the frequency of the exacerbations and symptomatology as well as other important outcomes such as the functional, respiratory capacity among others.

DETAILED DESCRIPTION:
The use of bronchodilators is an invaluable tool in COPD, in outcomes such as the exacerbation preventions, improvement of symptoms and exercise capacity and therefore in quality of life. However, as the efficacy as the security such as bronchodilators benefits that have only been characterized in patients with COPD secondary to smoking and it is only assumed benefits in COPD by other causes but without confirmation.

There are no national or international studies that describe the ultra long-acting bronchodilator's efficacy and security in COPD secondary to biomass exposure (BE).

The proportion of patients with COPD secondary by biomass exposure vary between 20-30%, depending on what kind of study and population, which is an important number leading to a great mortality, morbidity, social and economic, being important to characterize in a better way several relevant aspects such as the long period treatment response.

The proportion of patients with COPD by BE presents major proportion of phenotype "bronchitis" with major condition of peripheral airways level, with major proportion of dyspnoea and a decrease in the quality of life. It is precisely in these aspects where have been demonstrated benefits with ultra long-acting bronchodilators, as consequence, it is expected that this group of patients will be benefitted equal and perhaps in greater magnitude that those that are encompassed in the "emphysematous" phenotype.

Additionally, it is well described that the sub-diagnostic and sub-optimum treatment in patients with COPD in first level; because this kind of patients generally have low social-economic status and assuming that in the first level they will find the principal attention, it would be important to define major therapeutic alternatives in them.

As it was mentioned before, the exercising capacity is a functional outcome deeply studied with prognostic capacity in patients with COPD secondary to smoking; it is probably that it could be an outcome with major impact in this special group of patients (COPD secondary to biomass exposure), because they live, in general, in rural areas, heads of household and therefore, in terms of social rolls their functionality requirement is higher.

Finally, there is a finding well described the low adherence to patient's treatment with COPD, with various reasons including low economic resources and others such as devices of complicated application, multiple dosage, etc. Due to the fact that most of the people who suffer COPD by biomass exposure are women dedicated to housework all the day, it is probable that this kind of medicines (dosage once a day) as well as free treatment, is a strategy that improves the treatment adherence and could represent an improvement in the important outcomes in this devastating disease (functional capacity, quality of life, frequency of exacerbations, mortality).

ELIGIBILITY:
Inclusion Criteria:

1. Age: 50-80 years
2. Female (female eligibility criteria are: Women in no fertile age who are non pregnant and committed to use effective contraception).*See note.
3. Relation FEV1/FVC less than 70% of predicted and the index obtained by the relation between the hours and the years of exposure (IEHL) more than 100 hrs/year (COPD of any grade or symptomatic).
4. Be able to assist at all the study visits.
5. Informed consent signed.
6. Be able to perform the functional pulmonary test satisfactorily.
7. Without any contraindication to perform any functional pulmonary test or exercise ( six-minute walking test.
8. Stable COPD (No history of exacerbations in the last 6 weeks previous to the inclusion).
9. Smoking index less than 5.
10. If the subject is chronic - degenerative diseases associated, these must be controlled.
11. II-III functional class that allow her assist to the study visits.

    *Note: This problem predominates in WOMEN, as gender and roles (predominately in rural areas) who are the ones that cook and are exposed enough time to appear the comorbidity associated (COPD, headache, backache, conjunctival irritation, etc). That is why in this study were included only women because this is a problem of gender and poverty.
12. Women with at least 5 years with amenorrhea (postmenopause).

Exclusion Criteria:

1. History of:

   * Allergy or known intolerance to any of the bronchodilator drugs in the study.
   * Asthma, bronchiectasis (as tuberculosis, whooping cough or other infection sequelae associated in the clinic history), tuberculosis, COPD recent exacerbation or acute respiratory infection.
   * Cardiovascular disease recent (less than 3 months) that contraindicate the functional pulmonary test.
2. Patients of childbearing age who do not agree to use effective methods of contraception.
3. Patients with suspected cancer at any level.

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Changes in quality of life (Saint George Respiratory Questionnaire (SGRQ)) | Baseline, 1, 3 and 6 months
  Changes in quality of life with SGRQ score.

SECONDARY OUTCOMES:
Changes in quality of life (COPD Assessment Test (CAT) | Baseline, 1, 3 and 6 months
  Changes in quality of life with CAT score.
Changes in dyspnea (modified Medical Research Council (mMRC) score. | Baseline, 1, 3 and 6 months
  Changes in dyspnea by mMRC score
Changes in dyspnea (Baseline Dyspnea Index (BDI) and Transition Dyspnea Index (TDI) questionnaires). | Baseline, 1, 3 and 6 months
  Changes in dyspnea with BDI/TDI scores.
Changes in pulmonary function 1 (inspiratory capacity (IC)) | Baseline, 1, 3 and 6 months
  Changes in IC in mL
Changes in pulmonary function (forced respiratory volume in the first second (FEV1) | Baseline, 1, 3 and 6 months
  Changes in FEV1 in mL.
Changes on the pulmonary function in functional capacity (walked meters on six minute walking test, 6MWT) from baseline to 6 month treatment. | Baseline, 1, 3 and 6 months
  Changes on the pulmonary function in functional capacity

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra Ramírez-Venegas, M.Cs., Principal Investigator — Instituto Nacional de Enfermedades Respiratorias, "Ismael Cosío Villegas"
Locations (1):
- Instituto Nacional de Enfermedades Respiratorias, "Ismael Cosío Villegas", Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Bruce N, Perez-Padilla R, Albalak R. Indoor air pollution in developing countries: a major environmental and public health challenge. Bull World Health Organ. 2000;78(9):1078-92. PMID 11019457
- [Background] Torres-Duque C, Maldonado D, Perez-Padilla R, Ezzati M, Viegi G; Forum of International Respiratory Studies (FIRS) Task Force on Health Effects of Biomass Exposure. Biomass fuels and respiratory diseases: a review of the evidence. Proc Am Thorac Soc. 2008 Jul 15;5(5):577-90. doi: 10.1513/pats.200707-100RP. PMID 18625750
- [Background] Regalado J, Perez-Padilla R, Sansores R, Paramo Ramirez JI, Brauer M, Pare P, Vedal S. The effect of biomass burning on respiratory symptoms and lung function in rural Mexican women. Am J Respir Crit Care Med. 2006 Oct 15;174(8):901-5. doi: 10.1164/rccm.200503-479OC. Epub 2006 Jun 23. PMID 16799080
- [Background] Perez-Padilla R, Regalado J, Vedal S, Pare P, Chapela R, Sansores R, Selman M. Exposure to biomass smoke and chronic airway disease in Mexican women. A case-control study. Am J Respir Crit Care Med. 1996 Sep;154(3 Pt 1):701-6. doi: 10.1164/ajrccm.154.3.8810608.
- [Background] Barr RG, Bourbeau J, Camargo CA, Ram FS. Tiotropium for stable chronic obstructive pulmonary disease: A meta-analysis. Thorax. 2006 Oct;61(10):854-62. doi: 10.1136/thx.2006.063271. Epub 2006 Jul 14. PMID 16844726
- [Background] Tashkin DP, Celli B, Senn S, Burkhart D, Kesten S, Menjoge S, Decramer M; UPLIFT Study Investigators. A 4-year trial of tiotropium in chronic obstructive pulmonary disease. N Engl J Med. 2008 Oct 9;359(15):1543-54. doi: 10.1056/NEJMoa0805800. Epub 2008 Oct 5. PMID 18836213
- [Background] Donohue JF, van Noord JA, Bateman ED, Langley SJ, Lee A, Witek TJ Jr, Kesten S, Towse L. A 6-month, placebo-controlled study comparing lung function and health status changes in COPD patients treated with tiotropium or salmeterol. Chest. 2002 Jul;122(1):47-55. doi: 10.1378/chest.122.1.47. PMID 12114338
- [Background] Brusasco V, Hodder R, Miravitlles M, Korducki L, Towse L, Kesten S. Health outcomes following treatment for 6 months with once daily tiotropium compared with twice daily salmeterol in patients with COPD. Thorax. 2006 Jan;61(1):91. doi: 10.1136/thx.2005.brusascolett. No abstract available. PMID 16396956
- [Background] Vogelmeier C, Kardos P, Harari S, Gans SJ, Stenglein S, Thirlwell J. Formoterol mono- and combination therapy with tiotropium in patients with COPD: a 6-month study. Respir Med. 2008 Nov;102(11):1511-20. doi: 10.1016/j.rmed.2008.07.020. Epub 2008 Sep 19. PMID 18804362
- [Background] van Noord JA, Aumann JL, Janssens E, Smeets JJ, Verhaert J, Disse B, Mueller A, Cornelissen PJ. Comparison of tiotropium once daily, formoterol twice daily and both combined once daily in patients with COPD. Eur Respir J. 2005 Aug;26(2):214-22. doi: 10.1183/09031936.05.00140404. PMID 16055868
- [Background] Rennard S, Bantje T, Centanni S, Chanez P, Chuchalin A, D'Urzo A, Kornmann O, Perry S, Jack D, Owen R, Higgins M. A dose-ranging study of indacaterol in obstructive airways disease, with a tiotropium comparison. Respir Med. 2008 Jul;102(7):1033-44. doi: 10.1016/j.rmed.2008.02.001. Epub 2008 May 13. PMID 18479895
- [Background] Vogelmeier C, Hederer B, Glaab T, Schmidt H, Rutten-van Molken MP, Beeh KM, Rabe KF, Fabbri LM; POET-COPD Investigators. Tiotropium versus salmeterol for the prevention of exacerbations of COPD. N Engl J Med. 2011 Mar 24;364(12):1093-1103. doi: 10.1056/NEJMoa1008378. PMID 21428765
- [Background] Wedzicha JA, Seemungal TA. COPD exacerbations: defining their cause and prevention. Lancet. 2007 Sep 1;370(9589):786-96. doi: 10.1016/S0140-6736(07)61382-8. PMID 17765528
- [Background] Niewoehner DE, Rice K, Cote C, Paulson D, Cooper JA Jr, Korducki L, Cassino C, Kesten S. Prevention of exacerbations of chronic obstructive pulmonary disease with tiotropium, a once-daily inhaled anticholinergic bronchodilator: a randomized trial. Ann Intern Med. 2005 Sep 6;143(5):317-26. doi: 10.7326/0003-4819-143-5-200509060-00007. PMID 16144890
- [Background] Caballero A, Torres-Duque CA, Jaramillo C, Bolivar F, Sanabria F, Osorio P, Orduz C, Guevara DP, Maldonado D. Prevalence of COPD in five Colombian cities situated at low, medium, and high altitude (PREPOCOL study). Chest. 2008 Feb;133(2):343-9. doi: 10.1378/chest.07-1361. Epub 2007 Oct 20. PMID 17951621
- [Background] Menezes AM, Perez-Padilla R, Jardim JR, Muino A, Lopez MV, Valdivia G, Montes de Oca M, Talamo C, Hallal PC, Victora CG; PLATINO Team. Chronic obstructive pulmonary disease in five Latin American cities (the PLATINO study): a prevalence study. Lancet. 2005 Nov 26;366(9500):1875-81. doi: 10.1016/S0140-6736(05)67632-5. PMID 16310554
- [Background] Ramirez-Venegas A, Sansores RH, Perez-Padilla R, Regalado J, Velazquez A, Sanchez C, Mayar ME. Survival of patients with chronic obstructive pulmonary disease due to biomass smoke and tobacco. Am J Respir Crit Care Med. 2006 Feb 15;173(4):393-7. doi: 10.1164/rccm.200504-568OC. Epub 2005 Dec 1. PMID 16322646
- [Background] Aaron SD, Vandemheen KL, Fergusson D, Maltais F, Bourbeau J, Goldstein R, Balter M, O'Donnell D, McIvor A, Sharma S, Bishop G, Anthony J, Cowie R, Field S, Hirsch A, Hernandez P, Rivington R, Road J, Hoffstein V, Hodder R, Marciniuk D, McCormack D, Fox G, Cox G, Prins HB, Ford G, Bleskie D, Doucette S, Mayers I, Chapman K, Zamel N, FitzGerald M; Canadian Thoracic Society/Canadian Respiratory Clinical Research Consortium. Tiotropium in combination with placebo, salmeterol, or fluticasone-salmeterol for treatment of chronic obstructive pulmonary disease: a randomized trial. Ann Intern Med. 2007 Apr 17;146(8):545-55. doi: 10.7326/0003-4819-146-8-200704170-00152. Epub 2007 Feb 19. PMID 17310045
- [Background] Beier J, Chanez P, Martinot JB, Schreurs AJ, Tkacova R, Bao W, Jack D, Higgins M. Safety, tolerability and efficacy of indacaterol, a novel once-daily beta(2)-agonist, in patients with COPD: a 28-day randomised, placebo controlled clinical trial. Pulm Pharmacol Ther. 2007;20(6):740-9. doi: 10.1016/j.pupt.2006.09.001. Epub 2006 Sep 30. PMID 17088091
- [Background] Cazzola M, Ando F, Santus P, Ruggeri P, Di Marco F, Sanduzzi A, D'Amato M. A pilot study to assess the effects of combining fluticasone propionate/salmeterol and tiotropium on the airflow obstruction of patients with severe-to-very severe COPD. Pulm Pharmacol Ther. 2007;20(5):556-61. doi: 10.1016/j.pupt.2006.06.001. Epub 2006 Jul 7. PMID 16914336
- [Background] Fitzgerald MF, Fox JC. Emerging trends in the therapy of COPD: bronchodilators as mono- and combination therapies. Drug Discov Today. 2007 Jun;12(11-12):472-8. doi: 10.1016/j.drudis.2007.04.003. Epub 2007 Apr 26. PMID 17532532
- [Background] Wise RA, Tashkin DP. Optimizing treatment of chronic obstructive pulmonary disease: an assessment of current therapies. Am J Med. 2007 Aug;120(8 Suppl 1):S4-13. doi: 10.1016/j.amjmed.2007.04.007. PMID 17678942
- [Background] Vogelmeier C, Ramos-Barbon D, Jack D, Piggott S, Owen R, Higgins M, Kramer B; INTIME study investigators (INdacaterol & TIotropium: Measuring Efficacy). Indacaterol provides 24-hour bronchodilation in COPD: a placebo-controlled blinded comparison with tiotropium. Respir Res. 2010 Oct 5;11(1):135. doi: 10.1186/1465-9921-11-135. PMID 20920365
- [Background] Romieu I, Riojas-Rodriguez H, Marron-Mares AT, Schilmann A, Perez-Padilla R, Masera O. Improved biomass stove intervention in rural Mexico: impact on the respiratory health of women. Am J Respir Crit Care Med. 2009 Oct 1;180(7):649-56. doi: 10.1164/rccm.200810-1556OC. Epub 2009 Jun 25. PMID 19556519
- [Background] Julious SA, Campbell MJ. Tutorial in biostatistics: sample sizes for parallel group clinical trials with binary data. Stat Med. 2012 Oct 30;31(24):2904-36. doi: 10.1002/sim.5381. Epub 2012 Jun 19. PMID 22714646
- [Derived] Robles-Hernandez RE, Montiel-Lopez F, Velazquez-Uncal M, Sansores RH, Hernandez-Zenteno RJ, Perez-Padilla R, Ramirez-Venegas A. Efficacy of Indacaterol vs Tiotropium in COPD patients due to biomass exposure in improving quality of life and reducing symptoms. Respir Med. 2025 May;241:108074. doi: 10.1016/j.rmed.2025.108074. Epub 2025 Mar 30. PMID 40169096